CLINICAL TRIAL: NCT03099759
Title: Effectiveness of Various Vitamin D Protocols on Raising and Maintaining Blood Serum 25(OH)D3 Levels Over a Three Month Period
Brief Title: Vitamin D Raising and Maintaining Blood Serum 25(OH)D3 Levels
Acronym: VitD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Brentwood Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB 16-028
Record Dates: First submitted 2017-03-23; First posted 2017-04-04 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D Dosing Regimens; Blood Serum 25(OH)D3 Levels
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin Dose Group 100,000 Units (Active Comparator): 100,000 units Vitamin D2 one time only.
  Interventions: Dietary Supplement: Vitamin D
- Vitamin Dose Group 100,000 Units D2 (Active Comparator): 100,000 units vitamin D2 weekly for three months.
  Interventions: Dietary Supplement: Vitamin D
- Vitamin Dose Group 50,000/2,000 D2/D3 (Active Comparator): 50,000 units Vitamin D2 for 10 days followed by 2,000 units Vitamin D3 daily the remainder of the three month study period.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D2/D3
  Other Names: Ergocalciferol, cholecalciferol

SUMMARY:
Analyze the amount of change in blood serum Vitamin D levels in patients of 3 different dosing groups and how their levels change over a 3 month period of time.

DETAILED DESCRIPTION:
Vitamin D has shown multiple health benefits specifically in regards to bone healing. To the investigators knowledge there are currently no protocols for Vitamin D supplementation in the Orthopedic community for patients recovering from fractures. The investigators study will monitor 3 different groups of volunteers taking various Vitamin D regimens and how participants blood serum 25(OH)D3 levels are effected throughout a 3 month period. The 3 groups will include: 1) 100,000 units D2 once on day one, 2) 100,000 units D2 taken once a week x 12 weeks, 3) 50,000 units D2 x 10 days, then 2000 units D3 taken daily for the remainder of the study period. There will be 15-20 volunteers randomly assigned to each of the 3 groups. The investigators will have each volunteer from the 3 groups have blood drawn a total of 4 times throughout the course of this study: prior to the study, week 2, week 6, and week 12. From these results the investigators will determine which protocol most effectively raises and maintains vitamin D levels in the volunteers through this 3 month period. The investigators will also use this data to determine which protocol is not only most cost efficient but also easiest to follow by individuals. The investigators are hoping that this study may help finally develop a universal orthopedic protocol for vitamin D supplementation in patients recovering from fractures.

ELIGIBILITY:
Inclusion Criteria:

* Low Vitamin D level

Exclusion Criteria:

* Normal Vitamin D level, already taking Vitamin D, any form of steroids, weight-loss drugs, anti-tuberculosis drugs, high blood pressure drugs, high cholesterol drugs, endocrine disease, being treated for any form of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Vitamin D | Three Months
  Effectiveness of various Vitamin D protocols on raising and maintaining blood serum 25(OH)D3 levels over a three month period from baseline to 3 months with participants blood draws at initial, week 2, week 6 and week 12 time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Damien Billow, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No